CLINICAL TRIAL: NCT06873100
Title: Efficacy, Safety and Immunological Evaluation of Upadacitinib for Relapsing Polychondritis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, He Jing, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Upadacitinib RP
Record Dates: First submitted 2025-02-26; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-10

CONDITIONS: Relapsing Polychondritis
Keywords: Relapsing polychondritis; Upadacitinib
MeSH Terms: conditions — Polychondritis, Relapsing | interventions — upadacitinib; Adrenal Cortex Hormones; Immunosuppressive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Drug: Upadacitinib
- Countrol Group (Active Comparator)
  Interventions: Drug: corticosteroids and immunosuppressants

INTERVENTIONS:
Drug: Upadacitinib — Upadacitinib is an oral Janus kinase (JAK) inhibitor used in this study to treat patients with relapsing polychondritis. The drug is administered at a dose of 15 mg once daily for a duration of 24 weeks.
  Arms: Experimental Group
Drug: corticosteroids and immunosuppressants — Corticosteroids combined with immunosuppressants is a conventional treatment for relapsing polychondritis. In this study, it serves as the control arm against Upadacitinib for the treatment of relapsing polychondritis. Dosing is tailored to the individual patient's condition, with the selection of different types of corticosteroids and immunosuppressive agents based on the specific needs of the patient's clinical profile.
  Arms: Countrol Group

SUMMARY:
Relapsing polychondritis (RP) is a rare, systemic autoimmune disorder characterized by episodic inflammation of cartilaginous structures.

The goal of this clinical trial is to learn if drug Upadacitinib works to treat relapsing polychondritis in adults. It will also learn about the safety of drug Upadacitinib. The main questions it aims to answer are:

* Does drug Upadacitinib reduce the disease activity of relapsing polychondritis?
* What medical problems do participants have when taking drug Upadacitinib? Researchers will compare drug Upadacitinib to conventional therapies (treatment with corticosteroids combined with immunosuppressants) to see if drug Upadacitinib works to treat relapsing polychondritis.

Participants will:

* Take drug Upadacitinib or corticosteroids combined with immunosuppressants every day for 24 weeks.
* Visit the hospital once every month for checkups and tests. This clinical study will explore the efficacy and immunological evaluation of Upadacitinib in the treatment of RP.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female ≥18 and ≤70 years
* 2.Meet the revised Michet criteria
* 3.Patients had an inadequate response to standard treatment for ≥ 4 weeks. The background treatment included corticosteroids (≤0.5 mg/ kg), immunosuppressants ( methotrexate, hydroxychloroquine, azathioprine, mycophenolate mofetil leflunomide, or cyclophosphamide)
* 4. Negative urine pregnancy test
* 5. Written informed consent form

Exclusion Criteria:

Any subject who meets any of the following criteria shall be excluded:

* 1.Use rituximab or other monoclonal antibodies within 2 months.
* 2.1 months after treatment with high dose glucocorticoid (> 1 mg/kg/d).
* 3.Serious complications: heart failure (≥ New York Heart Association（NYHA） III grade), renal insufficiency (creatinine clearance rate ≤ 30 ml/min), liver function insufficiency (serum alanine transaminase or glutamic-pyruvic transaminaseT > 3 times normal upper limit, or total bilirubin > normal upper limit)
* 4.Other serious, progressive or uncontrollable hematological, gastrointestinal, endocrine, lung, heart, nerve, or brain diseases (including demyelination diseases, such as multiple sclerosis).
* 5.Known allergies, hyperresponsiveness or IL-2 or its excipients are intolerant.
* 6.Severe infections (including, but not limited to, hepatitis, pneumonia, bacteremia, pyelonephritis, Epstein-Barr virus, tuberculosis infection), hospitalization for infection, or intravenous antibiotics 2 months before the first dose of treatment.
* 7.Chest imaging showed abnormalities in malignant tumors or current active infections (including tuberculosis) within 3 months before the first use of the study.
* 8.Infected with HIV (HIV antibody positive serology) or hepatitis C (Hep C antibody positive serology). If seropositive, consult a doctor with expertise in the treatment of HIV or hepatitis C virus infection.
* 9.There has been any known malignant tumor or history of malignant tumor in the past 5 years (with the exception of non-melanoma skin cancer, non-melanoma skin cancer with no sign of recurrence or surgically cured cervical tumor within 3 months of use of the first study preparation).
* 10.There are uncontrolled mental or emotional disorders, including a history of drug and alcohol abuse over the past three years, which may hinder the successful completion of the study. 11.Within 3 months before the first injection of the research agent, during the study period or within 4 months after the last injection of the research agent, any live virus or bacterial vaccine is received or expected to be received. Bacillus Calmette-Guerin was vaccinated within 12 months after screening.
* 11.Pregnant and lactating women (WCBP) are reluctant to use medically approved contraceptives during and 12 months after treatment.
* 12.Men whose partners have fertility potential but do not want to use appropriate medically approved contraceptives during and within 12 months of treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CRP variation | 24 weeks
  Modification of inflammatory makers

SECONDARY OUTCOMES:
Relapsing Polychondritis Disease Activity Index | 24 weeks
Variation of lymphocyte subpopulations and cytokine during the treatment of upadacitinib | 24 weeks
  Cytokine and lymphocyte subgroups of T cell, B cell and NK cell are analyzed during the treatment.
Improvement of clinical symptom measured by 5-level EQ-5D version (EQ-5D-5L) | 24 weeks
  The EQ-5D-5L is a health-related quality-of-life instrument developed by the EuroQol Group. It is designed to measure health status across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.
Alteration of inflammatory biomarkers and pathways after treatment of upadacitinib | 24 weeks
  We will investigate the potential pathways through which Upadacitinib exerts its effects and examine the changes in inflammatory biomarkers during the experimental process
Incidence of Treatment-Emergent Adverse Events | 24 weeks
  Adverse events includes influenza-like symptoms, infection, fever, tumor,drug-induced liver and kidney damage.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Principal Investigator — Peking University Institute of Rheuamotology and Immunology
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China